CLINICAL TRIAL: NCT02281786
Title: A SINGLE-CENTER, RANDOMIZED, INVESTIGATOR/SUBJECT BLIND, SINGLE ASCENDING DOSE, PLACEBO CONTROLLED, PARALLEL STUDY TO INVESTIGATE THE SAFETY, TOLERABILITY AND PHARMACOKINETICS OF RO6926496 FOLLOWING INTRAVENOUS INFUSION IN HEALTHY SUBJECTS
Brief Title: A Study of RO6926496 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BP29462; 2014-003170-16 (EudraCT Number)
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Cohort 1 (Experimental): 8 volunteers (6 active, 2 placebo)
  Interventions: Drug: Placebo; Drug: RO6926496
- Cohort 2 (Experimental): 8 volunteers (6 active, 2 placebo)
  Interventions: Drug: Placebo; Drug: RO6926496
- Cohort 3 (Experimental): 8 volunteers (6 active, 2 placebo)
  Interventions: Drug: Placebo; Drug: RO6926496
- Cohort 4 (Experimental): 8 volunteers (6 active, 2 placebo)
  Interventions: Drug: Placebo; Drug: RO6926496
- Cohort 5 (Experimental): 8 volunteers (6 active, 2 placebo)
  Interventions: Drug: Placebo; Drug: RO6926496
- Cohort 6 (Experimental): 8 volunteers (6 active, 2 placebo)
  Interventions: Drug: Placebo; Drug: RO6926496

INTERVENTIONS:
Drug: Placebo — Matching placebo to RO6926496
Drug: RO6926496 — single, ascending dose, intravenous administration

SUMMARY:
This is a single center, randomized, investigator/subject blind, single ascending dose, placebo-controlled, parallel study that will evaluate the safety, tolerability and pharmacokinetics of RO6926496 in healthy male participants. The dose escalation is adaptive in nature. It is planned to enroll 48 subjects in 6 cohorts. The anticipated total duration of the study is 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants, 18 to 45 years of age; healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history
* A body mass index between 18 and 30 kg/m2
* Male subjects and their partners of childbearing potential must agree to use 2 methods of contraception, one of which must be a barrier method for the duration of the study

Exclusion Criteria:

* Positive hepatitis B, hepatitis C, or HIV infection
* History of any clinically significant disease or disorder
* Clinically significant abnormalities in laboratory test results
* Participation in an investigational drug or device study within 90 days prior to screening
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* History or presence of clinically significant ECG abnormalities
* Smokers who smoke more than 10 cigarettes daily or equivalent and unable or unwilling not to smoke during the in-clinic period
* Any clinically relevant history of hypersensitivity or allergic reactions
* Any familial history of early onset Alzheimer's disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 16 weeks

SECONDARY OUTCOMES:
Pharmacokinetic profile and parameters derived from serum concentrations of RO6926496 (composite outcome measure): area under the concentration-time curve (AUC), Cmax, tmax, clearance | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Leeds, United Kingdom